CLINICAL TRIAL: NCT00000381
Title: Fluoxetine for Anxious Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Boris Birmaher, MD, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH053681 (NIH); R01MH053681 (NIH); DSIR
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2005-12

CONDITIONS: Anxiety Disorders
Keywords: Adolescence; Anxiety Disorders; Child; Female; Fluoxetine; Male; Placebos; Serotonin Uptake Inhibitors; Anxiety Disorders -- *drug therapy; Fluoxetine -- *therapeutic use; Serotonin Uptake Inhibitors -- *therapeutic use
MeSH Terms: conditions — Anxiety Disorders | interventions — Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
The purpose of this study is to see if it is safe and effective to use fluoxetine to treat children and adolescents with Generalized Anxiety Disorder (GAD).

Anxiety disorders are one of the most common psychiatric disorders in children and adolescents, and can cause disturbances in the child's school, social, and family lives. Having an anxiety disorder puts a child at risk for depression and drug abuse, and appears to continue into adulthood. There is very little information on anxiety medications for children.

Children will be assigned randomly (like tossing a coin) to receive either fluoxetine or an inactive placebo for 12 weeks. Each child will be monitored for symptoms and side effects throughout the study. He/she will have blood tests at Weeks 4, 8, and 12 to measure drug levels in the blood. The study will last for 12 weeks.

A child is eligible for this study if he/she:

Is 8 to 17 years old and has anxiety disorder.

A child will not be eligible for this study if he/she:

Has current major depression, panic disorder, or obsessive-compulsive disorder, or abuses alcohol or drugs.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of fluoxetine as a treatment for children and adolescents with Generalized Anxiety Disorder (GAD).

Anxiety disorders are among the most common childhood and adolescent psychiatric disorders and are often associated with academic, social, and family morbidity. These disorders frequently increase the risk for developing other psychiatric disorders (e.g., depression, substance abuse), aggregate in families, and appear to continue into adulthood. Except for Obsessive-Compulsive Disorder, there are very few pharmacological treatment studies for childhood anxiety disorders. Given the sparsity and methodological problems of previous anxiety pharmacological studies, it is clear that further investigation of the use of pharmacological treatment of children and adolescents with these disorders is needed.

Patients are randomized to receive either fixed-dose fluoxetine or placebo for 12 weeks. Patients are assessed for psychiatric symptomatology, functional status, and side effects. In addition, to assess attainment of steady state and compliance with treatment, plasma levels of fluoxetine and norfluoxetine are measured at 4, 8, and 12 weeks. To standardize the treatment protocol and to assure that both groups (fluoxetine and placebo) receive equivalent nonpharmacological treatment, a manual is used. Potential predictors of clinical response (such as age, sex, duration and severity of anxiety, school absenteeism, sub-syndromal depressive symptoms, family history of anxiety or mood disorders) are explored.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Generalized anxiety disorder.

Exclusion Criteria:

-

Excluded:

Patients with current major depression, as well as patients with panic and obsessive-compulsive disorder.

-

Excluded:

Current substance abuse.

Ages: 8 Years to 17 Years | Sex: All
Age Groups: Child
Dates: Start 1997-06; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Birmaher, MD, Principal Investigator

REFERENCES:
- [Result] Birmaher B, Axelson DA, Monk K, Kalas C, Clark DB, Ehmann M, Bridge J, Heo J, Brent DA. Fluoxetine for the treatment of childhood anxiety disorders. J Am Acad Child Adolesc Psychiatry. 2003 Apr;42(4):415-23. doi: 10.1097/01.CHI.0000037049.04952.9F. PMID 12649628